CLINICAL TRIAL: NCT02982122
Title: A Randomized Clinical Trial Assessing the Effect of "Optimal" Cerebral Perfusion Pressure Monitoring in the Management of Severe Traumatic Brain Injury
Brief Title: CPPopt Guided Therapy: Assessment of Target Effectiveness
Acronym: COGITATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COGITATE
Record Dates: First submitted 2016-11-23; First posted 2016-12-05 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Brain Injuries, Traumatic; Cerebrovascular Circulation; Homeostasis
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Vasoconstrictor Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPPopt intervention group (Experimental): Patients are managed according to Brain Trauma Foundation guidelines, except for CPP where the CPPopt is targeted.
  Interventions: Other: For both groups, CPP targets will be achieved first by ICP control if this is raised and then by ABP support by titration (up or down) of vasopressors and fluids according to local protocols.
- CPP control group (Active Comparator): Patients are managed according to Brain Trauma Foundation guidelines with CPP between 60 and 70 mmHg.
  CPPopt information is recorded but hidden for the treating clinicians.
  Interventions: Other: For both groups, CPP targets will be achieved first by ICP control if this is raised and then by ABP support by titration (up or down) of vasopressors and fluids according to local protocols.

INTERVENTIONS:
Other: For both groups, CPP targets will be achieved first by ICP control if this is raised and then by ABP support by titration (up or down) of vasopressors and fluids according to local protocols. — For both groups, CPP targets will be achieved first by ICP control if this is raised and then by ABP support by titration (up or down) of vasopressors and fluids according to local protocols.

SUMMARY:
Despite improvements in management, mortality in severe traumatic brain injury (TBI) remains 25% and only 40% of patients survive without major handicap. Medical/surgical interventions aim to maintain adequate brain perfusion, which is critically dependent on cerebral perfusion pressure (CPP); calculated as the difference between mean arterial pressure (MAP) and intracranial pressure (ICP). Current guidelines aim for a CPP above 50 mmHg, based on population means. However, this 'one size fits all' approach is flawed, because the relation between CPP and brain perfusion varies between individuals. Further, this approach takes no account of autoregulation, a key protective mechanism that maintains cerebral perfusion despite CPP fluctuations.

Autoregulation is variably preserved following TBI, and there are large between patient variances in the 'optimal' CPP (CPPopt) at which autoregulation operates best. Individual CPPopt can be retrieved automatically by plotting autoregulation data against the CPP over a certain time window. The investigators have shown that maintenance of CPP close to CPPopt is associated with improved outcomes. These data pose the hypothesis that optimisation of management in individuals may be achieved by using the zone of optimal autoregulation as a basis for defining individualised CPP targets.

The investigators propose, together with collaborators in the CPPopt study group (Maastricht, Cambridge, Leuven and Aachen) to set up a pilot (multicenter) feasibility study to develop a protocol for a definitive outcome randomized controlled trial (RCT). This study aims to develop protocols for CPPopt guided critical care, and show that they maintain patients closer to their optimum perfusion levels than standard protocols which keep above a population CPP threshold of 60 mmHg.

Hence, the main objective is to offer clinicians monitoring and therapy algorithms that achieve individualized optimal CPPopt targets and potentially improve TBI outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any adult severe TBI patient requiring multimodality monitoring and ICP-directed therapy for at least 24 hrs on the assessment of the recruiting team.
* Start randomization within 24 hrs after ICU admission.
* Deferred informed consent or deferred proxy assent from relatives/legal representative (consultee).
* Exception for enrolling a patient past the 24 hour window: A patient who is admitted to the hospital and later experiences neuro-worsening that is not due to a systemic insult, (e.g. myocardial infarction, arrhythmia, pulmonary embolus, systemic hemorrhage) but due to a presumptive intracranial cause, and subsequently requires an ICP monitor, may be screened for enrolment. Consent, randomization, and monitor placement must be done within 48 hours from injury in order for the patient to qualify.

Exclusion Criteria:

* Patients < 18 years old.
* Known pregnancy.
* Moribund at presentation (e.g. bilaterally absent pupillary responses)
* Patients with primary decompressive craniectomy.
* Patients already enrolled in > 1 other research studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Percentage of monitoring time with measured CPP within 5 mmHg of calculated CPPopt | First 5 days during intensive care unit admission
  Main feasible endpoint: In pilot studies, we showed that, on average, patients spent a mean (+SD) of 30% ( 8%) of their monitored time with measured CPP within 5 mmHg of CPPopt. The study will be powered to target an increase in this metric to 50% of monitored time.

SECONDARY OUTCOMES:
Treatment Intensity Level (TIL) score | First 5 days during intensive care unit admission
  Main safety secondary endpoint: A change in daily TIL score of > 3 is representative of a clinical significant escalation of TBI treatment from basic ICP management to second tier therapies known to carry risk of harm and therefore is expected to represent a clinically significant potentially harmful effect of CPPopt guided management.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Roekaerts, professor, Study Chair — Maastricht University Medical Center
Locations (2):
- Academic Hospital Leuven, Leuven, Belgium
- The Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Result] Aries MJ, Wesselink R, Elting JW, Donnelly J, Czosnyka M, Ercole A, Maurits NM, Smielewski P. Enhanced Visualization of Optimal Cerebral Perfusion Pressure Over Time to Support Clinical Decision Making. Crit Care Med. 2016 Oct;44(10):e996-9. doi: 10.1097/CCM.0000000000001816. PMID 27270178
- [Result] Zuercher P, Groen JL, Aries MJ, Steyerberg EW, Maas AI, Ercole A, Menon DK. Reliability and Validity of the Therapy Intensity Level Scale: Analysis of Clinimetric Properties of a Novel Approach to Assess Management of Intracranial Pressure in Traumatic Brain Injury. J Neurotrauma. 2016 Oct 1;33(19):1768-1774. doi: 10.1089/neu.2015.4266. Epub 2016 Feb 11. PMID 26866876
- [Result] Donnelly J, Aries MJ, Czosnyka M. Further understanding of cerebral autoregulation at the bedside: possible implications for future therapy. Expert Rev Neurother. 2015 Feb;15(2):169-85. doi: 10.1586/14737175.2015.996552. PMID 25614952
- [Result] Aries MJ, Czosnyka M, Budohoski KP, Steiner LA, Lavinio A, Kolias AG, Hutchinson PJ, Brady KM, Menon DK, Pickard JD, Smielewski P. Continuous determination of optimal cerebral perfusion pressure in traumatic brain injury. Crit Care Med. 2012 Aug;40(8):2456-63. doi: 10.1097/CCM.0b013e3182514eb6. PMID 22622398
- [Derived] Beqiri E, Smielewski P, Robba C, Czosnyka M, Cabeleira MT, Tas J, Donnelly J, Outtrim JG, Hutchinson P, Menon D, Meyfroidt G, Depreitere B, Aries MJ, Ercole A. Feasibility of individualised severe traumatic brain injury management using an automated assessment of optimal cerebral perfusion pressure: the COGiTATE phase II study protocol. BMJ Open. 2019 Sep 20;9(9):e030727. doi: 10.1136/bmjopen-2019-030727. PMID 31542757